CLINICAL TRIAL: NCT04186273
Title: Post-operative Topical Administration of Fibrosis Inhibiting Compound FS2 in a Double-blind, Randomized, Vehicle-controlled Study Evaluating the Safety and Prevention of Cutaneous Scarring in Skin Grafts and Donor Sites.
Brief Title: Clinical Safety and Scar Prevention Study of a Topical Antifibrotic Compound FS2.
Acronym: FS2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Papp, Medical Director, BCPFF Burn Unit and Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H16-02491
Record Dates: First submitted 2019-11-15; First posted 2019-12-04 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Scar; Cicatrix; Hypertrophic Scar; Skin Graft Scar; Skin Graft Complications; Donor Site Complication; Keloid
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Intervention Model Description: QUADRUPLE-BLINDED, RANDOMIZED, VEHICLE-CONTROLLED STUDY INTRA-SUBJECT CONTROLS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PRINCIPLE INVESTIGATOR/ INVESTIGATORS/ SPONSOR/ OUTCOME ASSESSOR/ PATIENT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Donor Site Wound, Vehicle (Sham Comparator): A vehicle moisturizing cream base applied to a bisected area of the donor site wound (from where the skin graft skin harvested).
  Interventions: Other: Vehicle moisture balancing base
- Donor Site Wound, FS2 0.25 (Experimental): A moisturizing cream base containing 0.25%w/w of FS2, applied to a bisected area of the donor site wound (from where the skin graft skin harvested).
  Interventions: Drug: Fibrosis-Inhibiting-Compound-FS2
- Donor Site Wound, FS2 0.5 (Experimental): A moisturizing cream base containing 0.50%w/w of FS2, applied to a bisected area of the donor site wound (from where the skin graft skin harvested)
  Interventions: Drug: Fibrosis-Inhibiting-Compound-FS2
- Skin Graft Wound, Vehicle (Sham Comparator): A vehicle moisturizing cream base applied to a bisected area of the skin grafted wound site.
  Interventions: Other: Vehicle moisture balancing base
- Skin Graft Wound, FS2 0.25 (Experimental): A moisturizing cream base containing 0.25%w/w of FS2, applied to a bisected area of the skin grafted wound site.
  Interventions: Drug: Fibrosis-Inhibiting-Compound-FS2
- Skin Graft Wound, FS2 0.5 (Experimental): A moisturizing cream base containing 0.50%w/w of FS2, applied to a bisected area of the skin grafted wound site.
  Interventions: Drug: Fibrosis-Inhibiting-Compound-FS2

INTERVENTIONS:
Drug: Fibrosis-Inhibiting-Compound-FS2 — There are three (3) experimental interventions: vehicle moisture balancing base, FS2-0.25 moisturizer, and 0.5 moisturizing base.
  Other Names: FS2
  Arms: Donor Site Wound, FS2 0.25; Donor Site Wound, FS2 0.5; Skin Graft Wound, FS2 0.25; Skin Graft Wound, FS2 0.5
Other: Vehicle moisture balancing base — Vehicle base without FS2.
  Other Names: Vehicle
  Arms: Donor Site Wound, Vehicle; Skin Graft Wound, Vehicle

SUMMARY:
The study will investigate the safety and effectiveness of daily post surgical scar management, using a moisture-balancing base product containing different amounts of a novel (NCE) antifibrogenic compound FS2, a natural metabolite of the kynurenine pathway. Results of recent peer-reviewed, pre-clinical evidence warrant further investigation to validate therapeutic scar preventive efficacy of topically administered/delivered FS2. There are no known safety concerns with current product formulations. Recent Phase I clinical safety and tolerability data further support continuation of the research proposed in this study.

DETAILED DESCRIPTION:
Study Arms (Investigational Conditions):

Total of 6, categorized by type of wound and treatment allocation.

Description of Study Arms:

The quality of tissue repair and scarring will be evaluated in two different, bisected post-surgical sites on the same Participant. Each wound site represents a Study Arm. Each wound site will receive two treatments, one of which is always a vehicle. In total the two wound types provide a total of 6 Study Arms for statistical analysis.

Arm 1 / Wound Type 1 (skin grafted wounds: 3-treatment groups): The wound site (injury) that requires skin grafting surgery to remove normal, uninjured skin from the same Participant to cover and repair a deep wound (a "skin graft").

Arm 2 / Wound Type (donor skin graft harvest site; 3-treatment groups): A surgical wound where a piece of normal skin is removed at uniform depth using a dermatome to harvest a skin graft ("skin graft harvest site").

The bisected wound site is randomly assigned either a control or FS2 cream treatment.

Treatment Groups: Each wound site will be used to investigate and compare three different treatments. Participants will apply the investigated treatments ("IP") as directed to allocated bisected sections of the skin grafted wound and donor wound site for 90 days. Follow-on assessments will be conducted with additional study visits on Days 180 and 270 (study endpoint).

There are four (4) differently labelled products as follows:

Treatment-1 (IP1) A single, daily application of a moisturizing cream-base.

Treatment-2 (IP2) A single, daily application of a moisturizing cream-base with FS2 (0.50% w/w).

Treatment-3 (IP3) A single, daily application of a moisturizing cream-base with FS2 (0.25% w/w). IP3 will have two different product labels to conceal the identity of the vehicle.

Control-cream (IP1), and treatments IP2 and IP3 each containing 0.50%w/w or 0.25%w/w FS2 respectively, will be topically applied to designated treatment sites once per day for a period of 90 days. Investigator and participant will be blinded from both identity of treatment product and randomized location. Each participant will be provided a different cream for each bisected-site for a total of four (4) differently labelled creams; two for the donor site, and two for the skin grafted site. Participants will discuss and be informed/reminded at each visit about study design, responsibilities, possible adverse events, proper daily wound care and cream application methods.

ELIGIBILITY:
Inclusion Criteria:

1. Medically able to consent to study requirements
2. Adult, male and female trauma patients
3. Ages 18 to 65 years of age
4. Fluent in English (able to consent without a translator)
5. Isolated skin wound of 3% Total Body Surface Area
6. Participant requires partial thickness skin graft (meshed/non-meshed), face and genitalia excluded.
7. Grafted skin is between 100 cm2 and 600 cm2
8. Maximum skin graft expansion ratio is 1:1.5

Exclusion Criteria:

1. Medically unable to consent to study requirements
2. Require an English translator to lawfully consent to the study and its requirements
3. Treatment sights (skin graft sights) located on the face and genitalia
4. Expected to be medically unstable for the duration of the study period and an additional 1-month thereafter
5. Pregnant, or attempting to become pregnant
6. Known immunosuppression or immunosuppressive illness
7. Subjects who had taken part in a clinical trial within 3 months prior to admission to this trial or who are currently participating in a clinical trial, whether an investigational drug was used or not.
8. Subjects who had any clinical evidence of severe ongoing or prolonged depression or mental illness
9. Subjects who smoke more than 20 cigarettes a day
10. Subjects who demonstrated evidence of drug abuse
11. Any other diagnosis, condition, physical or geographical limitation with the participant that may render, or increases the likelihood of rendering, him/her unable to complete the entire study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) | 0-9 months
  Differences in clinical scale scoring of healing, complications and scar severity using Vancouver Scar Scale. Investigator assessment of target scar or keloid using the Vancouver Scar Scale (VSS). Scale parameters include: Pigmentation (0-2), Vascularity (0-3), Pliability (0-5), and Height (0-3). Scale measurements include: minimum score of 0 = normal to a maximum score of 2, 3 or 5 depending on the parameter measured.
Patient and Observer Scar Assessment Scale (POSAS) | 0-9 months
  Differences in clinical scale scoring of healing, complications and scar severity using Patient and Observer Scar Assessment Scale (POSAS). Investigator assessment of target scar or keloid using the Patient and Observer Scar Assessment Scale (POSAS). Scale parameters include: Vascularity, Pigmentation, Thickness, Relief, Pliability, and Surface Area. Scale measurements include: minimum score of 1 = normal skin to a maximum score of 10 = worst scar imaginable.

SECONDARY OUTCOMES:
Adverse Events | 0-9 months
  To evaluate and compare Treatment safety by the proportion of adverse events in each treatment arm.
Vital Signs - systolic blood pressure | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal systolic blood pressures in each participant.
Vital Signs - diastolic blood pressure | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal diastolic blood pressures in participant.
Vital Signs - Heart Rate | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal heart rates in each participant.
Vital Signs - Respiratory Rate | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal respiratory rates in each participant.
Vital Signs - Oral Temperature | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal temperatures in each participant.
Physical Exam Findings | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal physical exam findings in each participant.
Clinical Chemistry Results | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal clinical chemistry results in each participant.
Hematology Results | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal hematology results for each participant.
Urine Analysis Results | 0-9 months
  To evaluate and compare Treatment safety by the proportion of abnormal urine analysis results for each participant.
FS2 Pharmacokinetic urine analysis data | 0-2 hours; 0-9 months
  To obtain, evaluate and compare total urine drug concentrations for each participant and compare clearance normalized by estimated volume of distribution (Vd).
FS2 Pharmacokinetic blood analysis data | 0-2 hours; 0-9 months
  To obtain, evaluate and compare total blood drug concentrations for each participant and compare clearance normalized by estimated volume of distribution (Vd).
Pain Management | 0-9months
  Pain Visual Analog Scale longitudinal comparison of subjective changes for each participant.
  Pain, Visual analog scale (score 0-none to 10-worse)
Histology (Tissue Biopsies) | 3 months and 9 months
  Evaluate and compare pathological assessments of punch biopsies obtained from each treatment site and compare intra site subjective findings (qualitative) for each.
Histology (Tissue Biopsies) | 3 months and 9 months
  Evaluate and compare intra site scar elevation index ratios (comparative ratio of normal skin dimensions (e.g. thickness) to those of an adjacent scar). Assessment requires histology sections of punch biopsies obtained from each treatment site and further substantiates Outcome 16 above.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Papp, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- VGH Burn Unit, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to disseminate individual participant data at this time, beyond what will be accessible through publication.

REFERENCES:
- [Background] Papp A, Hartwell R, Evans M, Ghahary A. The Safety and Tolerability of Topically Delivered Kynurenic Acid in Humans. A Phase 1 Randomized Double-Blind Clinical Trial. J Pharm Sci. 2018 Jun;107(6):1572-1576. doi: 10.1016/j.xphs.2018.01.023. Epub 2018 Feb 6. PMID 29421218